CLINICAL TRIAL: NCT02481336
Title: Integrating Clinical and Genomic Profiles for Prediction and Prevention of Chemotherapy-induced Neuropathy Via Big Bio-Data Analytics
Brief Title: To Study the Individual Variants of Chemotherapy-Induced Neurotoxicity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-103-395
Record Dates: First submitted 2015-06-09; First posted 2015-06-25 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-04

CONDITIONS: Neurotoxicity Syndromes
Keywords: Chemotherapy; Peripheral Neuropathy
MeSH Terms: conditions — Neurotoxicity Syndromes; Peripheral Nervous System Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Sample Collection with DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer patients receiving chemotherapy: Stage I-IV ovarian cancer receiving chemotherapy Paclitaxel/Carboplatin
  Stage II-IV endometrial cancer receiving chemotherapy Paclitaxel/Carboplatin
  Stage III & high risk stage II colorectal cancer receiving chemotherapy with mFOLFOX
  1. Questionnaires
  2. Peripheral nervous system examination
  3. Whole Genome Sequence
  Interventions: Other: Questionnaires; Procedure: Peripheral nervous system examination; Genetic: Whole Genome Sequence

INTERVENTIONS:
Other: Questionnaires — EORTC CIPN20 and EQ-5D-3L
Procedure: Peripheral nervous system examination — nerve conduction velocity (NCV), quantitative sensory test (QST), and nerve excitability test (NET)
Genetic: Whole Genome Sequence — Genetic Test : 10 mL blood will be collected in Blood Sample Collection

SUMMARY:
To study the risk prediction of chemotherapy-induced peripheral neuropathy (CIPN) by the clinical bioinformatics and genomic profile.

DETAILED DESCRIPTION:
This is a prospective, observational, cohort study, monitoring the chemotherapy-induced peripheral neurotoxicity by traditional clinical scales, neurological examinations, and semi-quantitative assessments. Moreover, all the genetic changes will be analyzed by next generation sequencing and we will try to identify relevant variants in individuals who suffer from chemotherapy-induced neurotoxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed epithelial ovarian cancer, endometrial cancer or adenocarcinoma of colon or rectum
2. Pathological stage I~IV for ovarian cancer, stage II~IV endometrial cancer or stage III & high risk stage II for colorectal cancer
3. Scheduled to receive adjuvant Paclitaxel/Carboplatin for ovarian or endometrial cancer, or mFOLFOX6 for colorectal cancer
4. Age ≥ 20 years old
5. ECOG Performance status 0-1
6. Adequate organ function

   Bone marrow:

   Absolute neutrophil count (ANC) ≥ 1.5 x 109/L WBC ≥ 3.0 x 109/L Platelet count ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL

   Hepatic:

   Total bilirubin level ≤ 1.0 x UNL AST and ALT ≤ 3.0 x UNL

   Renal:

   Creatinine level ≤ 1.5 mg/dL in men, ≤1.4 mg/dL in women; or Estimated CCr ≥ 60 mL/min (CCr is estimated by Cockcroft-Gault formula, as appendix III).
7. Negative pregnancy test for women of childbearing potential only
8. Patient willing to provide blood sample for research purposes
9. Written informed consent

Exclusion Criteria:

1. Prior treatment with neurotoxic chemotherapy, such as oxaliplatin, cisplatin, carboplatin, taxanes or vinca alkaloids
2. Receiving chemotherapy within 6 months
3. History of allergy to 5-FU or LV
4. Pre-existing peripheral neuropathy of any grade
5. A family history of a genetic or familial neuropathy
6. Active uncontrolled infection
7. Significant medical diseases, such as unstable angina, acute or recent myocardial infarction (<6 months before enrollment), COPD with frequent exacerbation, uncontrolled hypertension, ore cent CVA (<6 months before enrollment)
8. Poor compliance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total 300 cancer patients will be enrolled in National Cheng Kung University Hospital from March, 2015 to March, 2017. The subjects are stage I-IV ovarian cancer patients receiving chemotherapy Paclitaxel/Carboplatin, stage II-IV endometrial cancer patients receiving chemotherapy Paclitaxel/Carboplatin, stage III & high risk stage II colorectal cancer patients receiving chemotherapy with mFOLFOX.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events occurring after chemotherapy based on genomic profiling | up to 2 years after chemotherapy

SECONDARY OUTCOMES:
Changes in quality-of-life measured by EORTC CIPN20 | up to 2 years after chemotherapy
Changes in quality-of-life measured by EQ-5D-3L | up to 2 years after chemotherapy
Change from Baseline in nerve conduction velocity (NCV) | up to 2 years after chemotherapy
Change from Baseline in quantitative sensory test (QST) | up to 2 years after chemotherapy
Change from Baseline in nerve excitability test (NET) | up to 2 years after chemotherapy
Relapse-free survival | up to 5 years after chemotherapy
Overall Survival | up to 5 years after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Ru Shen, PHD, Study Chair — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided